CLINICAL TRIAL: NCT06678776
Title: Endoscopic Anatomy of the Breast Fascia System: A Reverse Development Theory
Brief Title: Endoscopic Anatomy of the Breast Fascia System
Status: Recruiting | Type: Observational
Sponsor: Haiyan Li (Other)
Responsible Party: Sponsor-Investigator, Haiyan Li, chief physician, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Other Study IDs: 2024ZSLYEC-560
Record Dates: First submitted 2024-10-27; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Disease; Anatomy
MeSH Terms: conditions — Breast Diseases | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic Surgery: patients who underwent endoscopic breast surgery
  Interventions: Procedure: surgery
- Reduction Mammaplasty: patients who underwent reduction mammaplasty
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — Explore the relationship between breast fascia development and surgical processes by repeatedly observing surgical videos of endoscopic mastectomy and reduction mammaplasty.

SUMMARY:
This study will focus on two key theories: the development theory of the breast fascia system and the reverse development theory. The research findings indicate that breast development generally follows a growth pattern from anterior to posterior, and from central to peripheral regions. However, an intriguing phenomenon contradicting this developmental process was discovered through endoscopic mastectomy, which has not been previously discussed. Based on the aforementioned theoretical analysis, this study includes patients who underwent endoscopic and reduction mammaplasty in the Department of Breast Surgery in the Sixth Affiliated Hospital of Sun Yat-sen University. The investigators proposed the following research framework: firstly, comprehensively understanding the structure of the breast fascia and the sequence of breast development through endoscope and existing research; secondly, exploring the relationship between breast fascia development and surgical processes by repeatedly observing surgical videos of endoscopic mastectomy and reduction mammaplasty; lastly, proposing a reverse development theory for breast fascia based on these theories in order to provide standardized and procedural guidance for breast surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients who need mastectomy and patients who need breast reduction during the study period.

Exclusion Criteria:

* breast conserving surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients of Breast Surgery in the Sixth Affiliated Hospital of Sun Yat-sen University.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Identification of ligaments | 1 year
  The identification of ligaments primarily relies on the observation of membranous structures, and record the number of cases.

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The corresponding database has not been established yet.